CLINICAL TRIAL: NCT05941598
Title: Electroacupuncture to Prevent Chemotherapy-Related Cognitive Impairment in Patients With Breast Cancer
Brief Title: Electroacupuncture for Chemotherapy-Related Cognitive Impairment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Shiyan Yan, Principal Investigator, Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: YACU003
Record Dates: First submitted 2023-06-08; First posted 2023-07-12 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Chemotherapy-Related Cognitive Impairment
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture (Experimental): After skin disinfection, acupuncture needles will be inserted into the acupoints. All needles will be manipulated to achieve deqi. Then, an electroacupuncture apparatus will be connected. The stimulation parameters will be continuous wave, 2 Hz, and the current intensity will be adjusted according to the participant's comfort level.
  Interventions: Device: Electroacupuncture
- Sham acupuncture (Sham Comparator): After skin disinfection, acupuncture needles will be inserted into acupoints that are unrelated to the treated syndromes. The needles will be inserted to a depth of 3 to 5 mm, without any manipulation or deqi. Then, the electronic acupuncture apparatus will be connected, with a continuous wave of 2 Hz. However, the intensity of electrical stimulation will be set to a minimum level that participants can perceive, and the apparatus will be turned off after 30 seconds of stimulation.
  Interventions: Device: Sham acupuncture

INTERVENTIONS:
Device: Electroacupuncture — Participants in the electroacupuncture group will receive electroacupuncture twice a week, with each session lasting 30 minutes. The treatment will start one week before chemotherapy and continue throughout the chemotherapy period.
  Arms: Electroacupuncture
Device: Sham acupuncture — Participants in the sham acupuncture group will receive minimal acupuncture twice a week, with each session lasting 30 minutes. The treatment will start one week before chemotherapy and continue throughout the chemotherapy period.
  Arms: Sham acupuncture

SUMMARY:
The objective of this trial is to evaluate the effect of electroacupuncture compared to sham acupuncture in preventing CRCI among breast cancer patients scheduled to undergo chemotherapy.

DETAILED DESCRIPTION:
Participants will be randomized to receive either acupuncture or sham acupuncture treatment. Both treatments will be administered twice a week, starting one week before chemotherapy and continuing throughout the chemotherapy period. The study outcomes will be evaluated at three time points: baseline (before acupuncture and chemotherapy), during chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle). Each cycle typically lasts for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with stage I-III breast cancer
2. Scheduled to undergo chemotherapy
3. Aged between 18 and 75 years
4. MoCA score ≥ 26
5. Voluntary agreement to participate in the study and sign an informed consent

Exclusion Criteria:

1. Demonstrated tumor metastasis or recurrence
2. Had a prior history of chemotherapy
3. Reported a history of brain tumors, head trauma or stroke
4. Were diagnosed with cognitive function-impaired disorders, such as Alzheimer's disease
5. Were unable to cooperate with testing for any reasons
6. Had severe hepatic or renal insufficiency
7. Had hemorrhagic disorders, including von Willebrand disease, or were taking anticoagulant or antiplatelet medication
8. Had an implanted cardiac pacemaker
9. Had a history of alcohol abuse or drug addiction
10. Were participating in another interventional trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
The incidence of chemotherapy-related cognitive impairment (CRCI) at the end of chemotherapy | After chemotherapy (21 days after the last chemotherapy cycle). Each chemotherapy cycle typically lasts for 4 weeks.
  All participants will undergo neuropsychological assessments at baseline and after chemotherapy. CRCI is defined as two or more test scores at or below -1.5 standard deviations (SDs), or a single test score at or below -2.0 SDs from baseline to the end of chemotherapy.

SECONDARY OUTCOMES:
Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  FACT-Cog will be used to assess cognitive function and its impact on cancer patients.
Montreal Cognitive Assessment (MoCA) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  MoCA will be used to identify the presence of cognitive impairment.
Functional Assessment of Cancer Therapy-General (FACT-G) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  FACT-G will be used to measure the impact of cancer and its treatment on patients' overall well-being.
General Anxiety Disorder-7 (GAD-7) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  GAD-7 will be used to assess the frequency and severity of symptoms such as excessive worry, restlessness and difficulty in relaxing.
Patient Health Questionnaire-9 (PHQ-9) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  PHQ-9 will be used to assess the frequency and severity of several symptoms commonly associated with depression.
Insomnia Severity Index (ISI) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  ISI will be used to assess the severity of insomnia symptoms and their impact on an individual's daily functioning
Patient-Reported Outcomes version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) | During chemotherapy (one day before the third chemotherapy cycle), after chemotherapy (21 days after the last chemotherapy cycle).
  PRO-CTCAE is a tool used to document self-reported adverse events and their severity on a 5-point scale. In our trial, we plan to evaluate 12 symptoms selected from the original PRO-CTCAE scale, specifically decreased appetite, nausea, vomiting, heartburn, bloating, constipation, diarrhea, abdominal pain, insomnia, fatigue, headache, and dizziness.

OTHER OUTCOMES:
Treatment safety | Adverse events will be observed and recorded throughout the trial. The study duration will depend on the chemotherapy cycle of each participant, which may range from 4 months to 8 months.
  Incidence of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Shiyan Yan, PhD, Principal Investigator — Beijing University of Chinese Medicine